CLINICAL TRIAL: NCT02922491
Title: EFFECT OF VITAMIN E SUPPLEMENTATION IN METHYLATION AND MICRORNAS PROFILE IN ADULT WOMEN WITH OVERWEIGHT
Brief Title: Effect of Vitamin E Supplementation in Methylation and microRNAs Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Rafaella Cristhine Pordeus Luna, Master in nutritional sciences, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: FUParaíba1
Record Dates: First submitted 2016-09-17; First posted 2016-10-04 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2017-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Vitamin E; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): 400 mg Vitamin E of synthetic source
  1 once daily during 2 months
  Interventions: Dietary Supplement: vitamin E
- Group 2 (Experimental): 400 mg Vitamin E of natural source
  1 once daily during 2 months
  Interventions: Dietary Supplement: vitamin E
- Group control (Placebo Comparator): 400 mg of starch
  1 once daily during 2 months
  Interventions: Dietary Supplement: starch
- No intervention (No Intervention): Without intervention

INTERVENTIONS:
Dietary Supplement: vitamin E — daily intake of vitamin E
  Arms: Group 1; Group 2
Dietary Supplement: starch — daily intake of starch (control)
  Arms: Group control

SUMMARY:
It is a study of clinical and interventional character, in which individuals who participate in the intervention will be selected for convenience of the project database entitled "Second Cycle Diagnosis and Intervention Food Situation, Nutrition and Noncommunicable Disease More Prevalent Population of the city of João Pessoa / PB ". They will be invited to participate in the intervention female subjects, overweight or obese, aged 20 and 59 years. The selected individuals will be distributed randomly into four groups: receive daily supplementation of 01 capsules containing 400 mg of vitamin E synthetic source (Group 1); receive daily supplementation of 01 capsules containing 400 mg of natural source vitamin E (Group 2); receive daily supplementation of 01 placebo capsule (control group); and non-intervention group. Individuals of intervention groups will receive dietary plan respecting individual needs, in order to control weight during the 08 weeks period. The subjects of the group without intervention, did not follow a diet plan, nor did they take vitamin E or placebo capsules, and were asked to continue their current eating habits over the 8-week period This project aims to evaluate whether vitamin E supplementation may modify the methylation and microRNAs profile.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects;
* Persons aged between 20 and 59 years;
* Overweight or obese;

Exclusion Criteria:

* Individuals consumed alcohol and / or chronic smokers;
* Individuals who do not have preserved cognitive status;
* Individuals users of multivitamins and mineral supplements, appetite suppressants and steroids;
* Pregnant women.

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Comparison of methylation profile of DNA in overweight and obese women before and then intervention with vitamin E | two months
Comparison of microRNAs profile in overweight and obese women before and then intervention with vitamin E | two months

CONTACTS AND LOCATIONS:
Locations (1):
- Rafaella Cristhine Pordeus Luna, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luna RCP, Dos Santos Nunes MK, Monteiro MGCA, da Silva CSO, do Nascimento RAF, Lima RPA, Pimenta FCF, de Oliveira NFP, Persuhn DC, de Almeida ATC, da Silva Diniz A, Pissetti CW, Vianna RPT, de Lima Ferreira FEL, Rodrigues Goncalves MDC, de Carvalho Costa MJ. alpha-Tocopherol influences glycaemic control and miR-9-3 DNA methylation in overweight and obese women under an energy-restricted diet: a randomized, double-blind, exploratory, controlled clinical trial. Nutr Metab (Lond). 2018 Jul 11;15:49. doi: 10.1186/s12986-018-0286-7. eCollection 2018. PMID 30008789